CLINICAL TRIAL: NCT07236424
Title: Effectiveness of Short-term Supervised Group Exercise Therapy, Walking and Education on Mental Health, Quality of Life and Mobility in Elderly Residents of Nursing Homes
Brief Title: Effectiveness of Exercise, Walking, and Education on Mental Health, Mobility and Quality of Life in Elderly Residents of Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mostar (Other)
Responsible Party: Principal Investigator, Antonija Hrkać, Associate professor, University of Mostar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Studija V
Record Dates: First submitted 2025-11-15; First posted 2025-11-19 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Mental Health Care; Depression Anxiety Disorder; Quality of Life
Keywords: Mental Health; Depression; Anxiety; Quality of Life; Older Adults; Exercise Therapy; Physiotherapy; Walking
MeSH Terms: conditions — Psychological Well-Being; Depression; Anxiety Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 22 participants
  Interventions: Behavioral: Physiotherapy
- Control group (No Intervention): 20 participants

INTERVENTIONS:
Behavioral: Physiotherapy — 1. Exercise therapy - stretching and breathing exercises, stabilization exercises, mobility exercises, and balance and coordination exercises.
     The exercises will be performed in a standing and lying position, with the possibility of using aids - gymnastic ball and resistance bands. Implementation - three times a week for 40 minutes, for a total of four weeks.
  2. Walking activity - three times a week for half an hour.
  3. Education on optimal positions and movement in everyday life activities - at the beginning of the study in one session lasting 60 minutes.
  Arms: Intervention Group

SUMMARY:
Clinical Trial This clinical trial aims to determine the impact of physiotherapy interventions on mental health, quality of life, and spinal mobility in older adults. The physiotherapy intervention will consist of group exercise therapy (3 times a week, 40 minutes, 4 weeks in total), walking activities (3 times a week, 30 minutes, 4 weeks in total), and education on optimal positions and movements in daily activities (one session lasting 60 minutes)

The main questions it aims to answer are:

1. Are group exercise therapy and walking optimal for reducing symptoms of depression and anxiety and improving quality of life in older adults placed in nursing homes in a short period of time
2. Do physiotherapy interventions improve spinal mobility (anteflexion and extension)?

DETAILED DESCRIPTION:
Population ageing is a worldwide phenomenon resulting from increased living standards, improved healthcare, and decreased birth rates. The proportion of people aged 60 and over continues to grow and is expected to exceed two billion by 2050, with 80% of them living in developed countries.

Ageing is associated with a decline in physical and mental capacities, increased risk of chronic diseases, and social isolation, leading to higher healthcare and social costs. However, many of these challenges can be prevented or mitigated through timely interventions. Global health initiatives promote Healthy and Active Ageing, focusing on maintaining longevity, well-being, and quality of life. Physical activity and exercise therapy are the most effective interventions for promoting physical and mental health, highlighting the essential role of physiotherapy. Physiotherapists are well-positioned to promote healthy ageing due to their accessibility, cost-effectiveness, and expertise in managing a wide range of health conditions. Increasing evidence shows that physiotherapy not only enhances physical function but also contributes significantly to the mental well-being of older adults.

Recent systematic reviews with meta-analyses have reported positive effects of exercise therapy and physical activity on reducing depression, anxiety, and improving quality of life among older adults. An umbrella review reports high benefits of physical activity for improving symptoms of depression, anxiety, and distress across a wide range of adult populations, including the general population, people with diagnosed mental health disorders, and people with chronic disease. A systematic review with meta-analysis confirmed exercise as an effective treatment for anxiety. However, the heterogeneity of the included studies does not provide clearer information about the optimal exercise methods, as well as the necessary parameters and ways of implementing exercise therapy. In addition, individual studies show conflicting results on the effects of physical activity in nursing home residents; one reports benefits of a structured exercise program on depressive symptoms and quality of life, while another finds no significant improvement with supervised moderate aerobic and resistance training.

Thus, this study aim is to determine the optimal methods of exercise therapy and physical activity, as well as other parameters such as frequency, intensity, supervision, and method of implementation, in improving mental health and quality of life in elderly people in a nursing home.

ELIGIBILITY:
Inclusion Criteria:

* both sexes, aged ≥ 65 years, with an optimal level of functional and cognitive abilities necessary to perform the exercises and understand the measurement scales.

Exclusion Criteria:

* significant cognitive and neurological impairments, functionally immobile persons, and persons who refuse to participate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes
Enrollment: 44 (Actual)
Dates: Start 2025-11-20 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Depression and Anxiety | From enrollment to the end of treatment at 4 weeks
  Hospital Anxiety and Depression Scale (0=best, 21=worst)

SECONDARY OUTCOMES:
Self-reported measure of health | From enrollment to end of the treatment at 4 weeks
  The 36-Item Short Form Survey; Eight domains: Physical functioning, Role limitations due to physical health, Role limitations due to emotional problems, Energy/fatigue, Emotional well-being, Social functioning, Pain and General Health (0 - worst, 100 - best)
Range of motion of extension and flexion in the lumbar spine | From enrollment to the end of treatment at 4 weeks
  Goniometer (extension 0-40°, flexion 0-70°; higher score best)

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing home "Ministro", Žepče, Žepče, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Lok N, Lok S, Canbaz M. The effect of physical activity on depressive symptoms and quality of life among elderly nursing home residents: Randomized controlled trial. Arch Gerontol Geriatr. 2017 May-Jun;70:92-98. doi: 10.1016/j.archger.2017.01.008. Epub 2017 Jan 16. PMID 28110207
- [Background] Underwood M, Lamb SE, Eldridge S, Sheehan B, Slowther AM, Spencer A, Thorogood M, Atherton N, Bremner SA, Devine A, Diaz-Ordaz K, Ellard DR, Potter R, Spanjers K, Taylor SJ. Exercise for depression in elderly residents of care homes: a cluster-randomised controlled trial. Lancet. 2013 Jul 6;382(9886):41-9. doi: 10.1016/S0140-6736(13)60649-2. Epub 2013 May 2. PMID 23643112
- [Background] Noetel M, Sanders T, Gallardo-Gomez D, Taylor P, Del Pozo Cruz B, van den Hoek D, Smith JJ, Mahoney J, Spathis J, Moresi M, Pagano R, Pagano L, Vasconcellos R, Arnott H, Varley B, Parker P, Biddle S, Lonsdale C. Effect of exercise for depression: systematic review and network meta-analysis of randomised controlled trials. BMJ. 2024 Feb 14;384:e075847. doi: 10.1136/bmj-2023-075847. PMID 38355154
- [Background] Singh B, Olds T, Curtis R, Dumuid D, Virgara R, Watson A, Szeto K, O'Connor E, Ferguson T, Eglitis E, Miatke A, Simpson CE, Maher C. Effectiveness of physical activity interventions for improving depression, anxiety and distress: an overview of systematic reviews. Br J Sports Med. 2023 Sep;57(18):1203-1209. doi: 10.1136/bjsports-2022-106195. Epub 2023 Feb 16. PMID 36796860
- [Background] Liu-Ambrose T, Li LC. Physiotherapy for Healthy Aging. Physiother Can. 2022 Jan 1;74(1):1-3. doi: 10.3138/ptc-2021-0106-gee. Epub 2022 Jan 31. No abstract available. PMID 35185240
- [Background] Rivadeneira MF, Mendieta MJ, Villavicencio J, Caicedo-Gallardo J, Buendia P. A multidimensional model of healthy ageing: proposal and evaluation of determinants based on a population survey in Ecuador. BMC Geriatr. 2021 Nov 1;21(1):615. doi: 10.1186/s12877-021-02548-5. PMID 34719380
- [Background] Johnston MC, Crilly M, Black C, Prescott GJ, Mercer SW. Defining and measuring multimorbidity: a systematic review of systematic reviews. Eur J Public Health. 2019 Feb 1;29(1):182-189. doi: 10.1093/eurpub/cky098. PMID 29878097